CLINICAL TRIAL: NCT06274983
Title: Investigating the Viability and Acceptability of an Interactive Virtual Reality (IVR) System on Physiotherapy Rehabilitation in Paediatric Duchenne Muscular Dystrophy (DMD) Patients
Brief Title: DMD- Interactive Virtual Reality Study
Acronym: DMD-IVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Sheffield Hallam University (Other); UCL Great Ormond Street Institute of Child Health (Other); Leeds General Infirmary (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH-2629
Record Dates: First submitted 2023-06-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2023-06

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IVR platform trial (Other): 8 DMD patients from Sheffield Children's Hospital and 8 DMD patients from Leeds Teaching Hospital to trial the IVR platform.
  Interventions: Device: IVR platform trial

INTERVENTIONS:
Device: IVR platform trial — 8 DMD patients from Sheffield Children's Hospital and 8 DMD patients from Leeds Teaching Hospital to trial the IVR platform. Patients will receive device training and then use the VR device at home for 12 weeks. Physiotherapists will conduct pre (visit 1) and post (visit 2) assessments to assess changes using a Goniometer (measures ankle range of movement), PEDSQL quality of life data, GAD-7 anxiety questions and the NorthStar Ambulatory Assessment.

SUMMARY:
This study will help determine if an Interactive Virtual Reality system can improve the physiotherapy of young patients with Duchenne muscular dystrophy (DMD).

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a genetic disease causing muscle weakness and wasting affecting 2,500 people in the UK. International Standards of Care recommend that children with DMD undertake a daily stretching programme to maintain maximum muscle extensibility and optimise function. A lot of children are not motivated to perform these exercises, leading to earlier complications, reduced function and a poorer long-term prognosis.

Our collaborative research group has previously developed an interactive Immersive Virtual Reality (IVR) system to improve the delivery, engagement and success of physiotherapy for adult amputees, burns' patients and children with upper limb injuries. VR headsets have become more accessible in terms of price, usability and portability.

In a recent PPI survey, 78% of paediatric DMD patients stated that a VR system could improve physiotherapy engagement and performance. This study will investigate the feasibility and acceptability of an IVR device on paediatric DMD rehabilitation.

In phase 1 of this study, clinicians, physiotherapists, parents, carers and patients will participate in a co-design workshop to explore core VR rehabilitation scenarios. An IVR platform will be developed that will emulate current DMD physiotherapy. In phase 2, investigators will ask therapists and children to take part in testing the IVR platform. VR scenarios will be further developed and then tested in a trial with 16 DMD patients aged 5-10 years.

Pre and post-trial assessments will be performed to determine the effect of the IVR system on improving physiotherapy adherence, muscle strength testing, quality of life and anxiety. Qualitative interviews and questionnaires will be conducted with patients and clinical staff to obtain feedback on patient acceptability as well as practicality and acceptability of using IVR in a clinical setting.

This study will help determine if an IVR system can improve the physiotherapy of young patients with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-10 years
* Diagnosed with Duchenne muscular dystrophy (DMD) and receiving lower limb physiotherapy care
* Ambulant patients
* Able to speak/understand English

Exclusion Criteria:

* Physical or cognitive difficulties indicating the child would struggle to use the device or complete study activities.
* Outside age range.
* Non-ambulant patients.
* Facial injuries precluding the use of HMD.
* Issues relating to balance that could be affected by VR.
* Severe visual impairment.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Compliance: Ratings of frequency of the DMD-IVR device use for the participant's to complete recommended physiotherapy exercises. | 8 weeks
  The physiotherapy team prescribe a defined frequency for use individualised for each child.
  Pre and Post Home diary: Families will be asked to complete a paper/electronic diary to capture compliance with current physio regime (including frequency of stretching and other activities for a 4 week 'pre intervention' period).
  The system will log the frequency of use of the DMD-VR platform during the 8 weeks (quantitative) which will be cross referenced with the patient completed activity diary.
Compliance: Ratings of duration of the DMD-IVR device use for the participant's to complete recommended physiotherapy exercises. | 8 weeks
  The physiotherapy team prescribe a defined time for use individualised for each child.
  Pre and Post Home diary: Families will be asked to complete a paper/electronic diary to capture compliance with current physio regime (including duration of stretching and other activities for a 4 week 'pre intervention' period).
  The system will log the duration of use of the DMD-VR platform during the 8 weeks (quantitative) which will be cross referenced with the patient completed activity diary.
Post-trial qualitative interviews on perceptions, acceptability, usability and effectiveness of DMD-IVR device in the context of the family's overall burden of care | 30 minutes
  A semi-structured interview will be conducted by the research nurse in person/phone with the patient and parent after the DMD-IVR rehabilitation at home trial (8 week). Open-ended questions provided qualitative data relating to acceptability, practicality, difficulty, pain and enjoyability, and participant attitudes towards the IVR system and its future deployment.
  Another semi-structured interview was conducted with the clinical staff by the researcher in person at the end of the trial to explore her attitudes towards the DMD-IVR device and future deployment (8 week).
  Both interviews were recorded, transcribed and anonymised.
DMD-IVR Effectiveness standard functional assessments: North Star Ambulatory Assessment (NSAA) | 10 minutes
  NSAA is a 17-item rating scale used to measure functional motor abilities in ambulant children with DMD.
  The test must be completed without the use of any thoracic brace or leg orthoses. Therapist asks the patient to complete activities listed below.
  The activities are graded as follows:
  2 - "Normal" - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another
  0 - Unable to achieve independently
  This scale is ordinal with 34 as the maximum score indicating fully-independent function. Several studies have shown that NSAA is a quick, specific, reliable, valid, and clinically relevant method to measure the functional motor ability of ambulant children with DMD. NSAA is considered to be suitable to be used in research and in a multicentric setting provided that adequate training is given. [https://www.physio-pedia.com/North_Star_Ambulatory_Assessment]
  Evaluation at the baseline
DMD-IVR effectiveness measures with a Timed test 4 stair climb | 10 minutes
  Evaluation at the baseline screening visit by the physiotherapist and at the end of the study (week 8).
DMD-IVR effectiveness measured joint range of movement using Goniometer (Standard BASELINE® 12-inch) | 10 minutes
  Goniometer device (Standard BASELINE® 12-inch plastic goniometer, (Model 12- 1000-Fabrication Enter- prises, Inc: White Plains, New York) will be use by the clinical staff before and after the patient's rehabilitation to document the initial and subsequent range of motion, evaluate their progress and to determine the level of disability. Clinical staff used the goniometer. To assess any changes in range of movement using goniometer measured ankle range of movement, plus any other joint range of movement physiotherapist deemed clinically valuable. The clinical team examined the differences between a range of movements join (flexion, extension, abduction, and adduction) before and after the VR rehabilitation. The greater the range of movement the better. Evaluation at the baseline screening visit by the physiotherapist and at the end of the study (week 8).

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Childrens NHS FT, Sheffield, South Yorkshire, United Kingdom